CLINICAL TRIAL: NCT05979857
Title: A Phase 1, Open-label, Multicenter, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SP-3164 in Patients With Relapsed/Refractory Non-Hodgkin's Lymphoma
Brief Title: Study of SP-3164 in Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Salarius Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SALA-003-NHL
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Lymphoma, Non-Hodgkin's, Adult
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Intervention Model Description: This study is a phase 1, open-label, multicenter, dose escalation (part 1) and dose selection optimization (part 2) study of SP-3164 in patients with R/R B-cell NHL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): For part 1 dose escalation, one patient per dose cohort will be initially recruited (accelerated titration dose-escalation, single-patient cohorts/dose level) for the first two dose levels or until the first instance of a ≥ Grade 2 toxicity (excluding Grade 2 neutropenia and lymphopenia and adverse events unequivocally due to the underlying disease or to an extraneous cause), or dose-limiting toxicity (DLT), whichever occurs earlier. Further cohorts will be recruited in blocks of three patients, i.e., 3+3 dose escalation design.
  Interventions: Drug: SP-3164
- Dose Optimization (Experimental): For part 2 dose selection optimization, two dose levels will be selected by the Safety Review Committee (SRC) based on review of all available data on safety, tolerability, PK, PD, and preliminary efficacy from part 1. The dose selection optimization will include only patients with R/R DLBCL and will randomize 1:1 approximately 30 new patients at the two selected dose levels (15 patients to each of the two selected dose levels) before declaring the RP2D. Assessment of PK/PD of SP-3164 will be included in part 2 dose selection optimization.
  Interventions: Drug: SP-3164

INTERVENTIONS:
Drug: SP-3164 — SP-3164, an oral next generation cereblon-binding molecular glue 'protein degrader'

SUMMARY:
The purpose of this research is to help researchers find out if SP-3164 is safe and if it may be of benefit in the treatment of patients with Non-Hodgkin's lymphoma that has progressed after prior treatment, or that never responded to previous treatment.

DETAILED DESCRIPTION:
SALA-003-NHL is a phase 1 open-label, multicenter, first-in-human study of SP-3164 in patients with R/R B-cell NHL that will be conducted in two parts. Part 1 is a dose escalation using a sequential accelerated titration design for the first two dose levels followed by a 3+3 dose escalation design to assess the safety and tolerability of SP-3164 in patients with R/R B-cell NHL. Upon completion of the dose escalation design and review of all available safety, tolerability, PK, PD, and preliminary efficacy data the Safety Review Committee (SRC) will recommend two dose levels for the randomized dose selection optimization (Part 2). The dose selection optimization will randomize 1:1 approximately 30 patients with R/R DLBCL to the two selected dose levels (15 new patients per dose level) to determine the recommended phase 2 dose (RP2D) and further characterize safety, tolerability, PK, PD, and preliminary efficacy data of SP-3164. SP-3164 will be administered orally once daily under fasting conditions on 7 consecutive on-treatment days followed by 7 consecutive off-treatment days. One treatment cycle will be defined as 28 days.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis (WHO 2016 criteria) of R/R B-cell NHL in dose escalation (part 1) and limited to R/R DLBCL in dose selection optimization (part 2) confirmed by biopsy and immunophenotyping

Dose escalation: at time of enrollment, R/R B-cell NHL patients per WHO 2016 criteria including DLBCL (including low grade transformed lymphoma), mantle cell lymphoma, follicular lymphoma, and marginal zone lymphoma and must:

* require treatment in the opinion of the Investigator
* received at least 2 lines of systemic therapy for B-cell NHL

Dose selection optimization: at time of enrollment, R/R DLBCL (including low grade transformed lymphoma) patients must have received 2 or 3 lines of systemic therapy for DLBCL

o Prior immunomodulatory imide drug (IMiD) therapy is allowed (e.g., lenalidomide)

Measurable disease per the 2017 International Working Group Consensus Response Evaluation Criteria for Lymphoma

Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1

Existing archival tumor tissue (fresh frozen paraffin embedded [FFPE], 5 unstained slides) not older than 2 years from Cycle 1 Day 1 or willingness to provide fresh tumor biopsy during screening

Normal organ and marrow function, defined by specific laboratory parameters

Ability to take orally administered medication

Washout period prior to Cycle 1 Day 1 of SP-3164: at least 21 days or 5 half-lives (whichever is shorter) from prior systemic anticancer treatment, including chemotherapy, biologic therapy, small molecule inhibitors, monoclonal antibodies, and any investigational agents; at least 14 days from palliative radiotherapy if ≤ 10 fractions or total dose ≤ 30 gray (Gy) or at least 28 days from radiotherapy if total dose > 30 Gy; at least 21 days from major surgery

Life expectancy of at least 3 months

Exclusion Criteria:

Patients with chronic lymphocytic leukemia, high grade B-cell lymphoma, or Richter's syndrome

Patients who have not recovered to Grade 1 toxicity or baseline due to any previous anticancer therapy according to the NCI CTCAE v5.0, excluding Grade 2 alopecia. Lymphopenia ≤ Grade 2 is allowed

Patients with primary central nervous system (CNS) lymphoma or active CNS or meningeal lymphomatous involvement

Persistent diarrhea or malabsorption of ≥ Grade 2 despite medical management

Impaired cardiac function or clinically significant cardiac disease, including symptomatic congestive heart failure, left ventricular ejection fraction (LVEF) < 50%, unstable angina pectoris or cardiac arrhythmias, baseline QTc (Fridericia) > 450 milliseconds, long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, myocardial infarct within 6 months of study enrollment, clinically significant pericardial disease

Solid organ transplant recipient

Allogeneic stem cell transplantation (SCT) recipient

Autologous SCT recipient <100 days from Cycle 1 Day 1 or otherwise not fully recovered from SCT-related toxicity

Completion of CAR-T therapy < 90 days from Cycle 1 Day 1

Systemic immunosuppressants and chronic systemic corticosteroids (at doses ≥ 10 mg/day of prednisone or equivalent) are prohibited

Malignant disease, other than that being treated in this study. Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) who have undergone potentially curative therapy are not excluded. Other exceptions include malignancies that were treated curatively and have not recurred within 3 years prior to Cycle 1 Day 1 and any malignancy considered indolent and that has never required therapy

Other concurrent severe or uncontrolled concomitant medical conditions that might cause unacceptable safety risks or compromise compliance with the protocol

Pregnant and breastfeeding women

Known history of HIV-positivity; known hepatitis B or hepatitis C virus infection

Men and women of child-bearing potential unwilling to use adequate contraception according to study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Characterize the Safety of SP-3164 | 4 months
  Dose Escalation (Part 1)
  • To characterize the safety, dose limiting toxicities (DLTs), and maximum tolerated dose (MTD) of SP-3164
Dose Escalation: Assess Dose Limiting Toxicities of SP-3164 | 6 months
  Dose Escalation (Part 1)
  • To characterize the safety, dose limiting toxicities (DLTs), and maximum tolerated dose (MTD) of SP-3164
Dose Escalation: Assess the Maximum Tolerated Dose of SP-3164 | 6 months
  Dose Escalation (Part 1)
  • To characterize the safety, dose limiting toxicities (DLTs), and maximum tolerated dose (MTD) of SP-3164
Dose Optimization: Further characterize the safety of the 2 selected doses of SP-3164 from Part 1 (dose escalation) | 6 months
  Dose Selection Optimization (Part 2)
  • To further characterize the safety of the two selected doses of SP-3164 from part 1 and determine the recommended phase 2 dose (RP2D) of SP-3164 for future studies
Dose Optimization: Determine the recommended phase 2 dose of SP-3164 for future studies | 6 months
  • To further characterize the safety of the two selected doses of SP-3164 from part 1 and determine the recommended phase 2 dose (RP2D) of SP-3164 for future studies

IPD SHARING:
Plan to Share IPD: No